CLINICAL TRIAL: NCT00275197
Title: An Eight-Week, Double-Blind, Group-Sequential Design, Placebo Controlled Trial To Evaluate The Safety And Efficacy Of The Co- Administration Of Sertraline And Elzasonan (CP-448,187) In Outpatients With Major Depressive Disorder
Brief Title: A Research Study to Compare the Treatments of a Combination of Elzasonan With Zoloft, to Zoloft Alone, or Placebo in People With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A7571001
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2008-11-03 (Estimated); Status verified 2008-10

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline

INTERVENTIONS:
Drug: Sertraline and Elzasonan Combination
Drug: Sertraline
Drug: Placebo

SUMMARY:
The major purpose of the study is to help determine whether giving the combination of Elzasonan with Zoloft to people with depression is a better treatment than taking Zoloft alone. This study will also compare the safety and tolerability of Elzasonan and Zoloft combination to Zoloft alone or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, 18 years of age or older with a diagnosis of recurrent, moderate-to-severe MDD without psychotic features (DSM-IV 296.3x, with a HAMD17 score >= to 22 and CGI-S >=4.
* MDD must be the primary psychiatric disorder that motivated the subject to seek treatment and the current episode must be at least 1 month in duration but no longer than 6 months in duration.

Exclusion Criteria:

* Subjects who, in the investigator's judgement, would require treatment with electroconvulsive therapy (ECT), or antipsychotics, or would require a change in intensity of psychotherapy, or subjects who would require treatment with any other psychotherapeutic drugs during the course of the trial.
* Subjects who have ever been diagnosed with Panic Disorder, Post-Traumatic Stress Disorder, Obsessive-Compulsive Disorder, Bipolar Affective Disorder, Schizophrenia, Schizoaffective Disorder or othe Psychotic Disorder, MDD with a seasonal pattern, or Dissociative Disorders per DSM-IV criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2005-12; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The estimated treatment difference (elzasonan plus sertraline - sertraline monotherapy) in MADRS (Montgomery-Asberg Depression Rating Scale) remission rates at Week 8 in patients with MDD.

SECONDARY OUTCOMES:
Change from baseline in: MADRS, CGI-I, CGI-S, HAMA, HAMD17, CSFQ, SOS-10 and PGID-D total scores at Week 8. Treatment differences in MADRS response rates at Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (4):
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Norwich, Connecticut
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Beachwood, Ohio
- Pfizer Investigational Site, Santiago, RM, Chile
- Estonia (3):
  - Pfizer Investigational Site, Viljandi, Viljandi Mk.
  - Pfizer Investigational Site, Pärnu
  - Pfizer Investigational Site, Tallinn
- Russia (5):
  - Pfizer Investigational Site, Gatchina, Leningradskaya Oblast'
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Rostov-on-Don
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Smolensk

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7571001&StudyName=A%20research%20study%20to%20compare%20the%20treatments%20of%20a%20combination%20of%20Elzasonan%20with%20Zoloft%2C%20to%20Zoloft%20alone%2C%20or%20placebo%20in%20people%20with